CLINICAL TRIAL: NCT00280475
Title: Randomized Phase III Trial of Postoperative Whole Brain Radiation Therapy Compared With Salvage Stereotactic Radiosurgery in Patients With One to Four Brain Metastasis: Japan Clinical Oncology Group Study (JCOG 0504)
Brief Title: A Trial of Postoperative Whole Brain Radiation Therapy vs. Salvage Stereotactic Radiosurgery Therapy for Metastasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haruhiko Fukuda (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor-Investigator, Haruhiko Fukuda, JCOG Data Center, Japan Clinical Oncology Group
Organization: Japan Clinical Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG0504; C000000307 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Brain Neoplasms; Neoplasm Metastasis
Keywords: Randomized Controlled Trials; Brain Neoplasms/Secondary; Brain Neoplasms/Radiotherapy; Radiosurgery
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Device: Whole brain radiation therapy arm
  Interventions: Device: Whole brain radiation therapy arm
- 2 (Experimental): Device: Salvage stereotactic radiosurgery arm
  Interventions: Device: Salvage stereotactic radiosurgery arm

INTERVENTIONS:
Device: Whole brain radiation therapy arm — Whole brain radiation therapy arm
  Arms: 1
Device: Salvage stereotactic radiosurgery arm — Salvage stereotactic radiosurgery arm
  Arms: 2

SUMMARY:
The aim of this study is to evaluate non-inferiority of salvage stereotactic radiosurgery (SRS) in the patients who received surgical resection for brain metastases in comparison with postoperative whole brain radiation therapy (WBRT).

DETAILED DESCRIPTION:
A randomized phase III study is started in Japan to compare postoperative whole brain radiation therapy with salvage stereotactic radiosurgery in patient with one to four brain metastases from lung, breast, and colorectal cancer.

Total of 270 patients will be accrued for this study from 21 institutions within three years. The primary endpoint is overall survival. The secondary endpoints are proportion of performance status (PS) preservation, proportion of mini-mental status examination (MMSE) preservation, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. one to four brain metastases with a maximum diameter of 3 cm or more for the largest lesion and additional lesions not exceeding 3 cm in diameter
2. all brain metastases localized within cerebrum or cerebellum
3. before surgical resection for brain metastasis, PS is 0-2, or 3 by cerebral nerve compression neurological deficits
4. surgical resection for the largest brain metastases has achieved
5. after surgical resection, four or fewer (0-4) residual lesions with maximum diameter under 3 cm
6. histologically proven non-small cell carcinoma, breast cancer or colorectal cancer
7. primary lesion and the other metastases (i.e. lung, liver, bone metastases except for brain) is consider to be controlled
8. an age of 20-79 years
9. no prior surgery or irradiation for brain
10. adequate organ function
11. written informed consent(If signing in consent form is difficult for the patient due to paralysis, signing by the family in place of the patient is permitted)

Exclusion Criteria:

1. synchronous or metachronous (within 5 years) malignancy other than carcinoma in situ or mucosal cancer
2. pregnant or breast-feeding women
3. severe mental disease
4. allergic to gadolinium contained contrast agents

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2006-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
overall survival | During the study conduct

SECONDARY OUTCOMES:
proportion of performance status (PS) preservation | During the study conduct
proportion of mini-mental status examination (MMSE) preservation | During the study conduct
adverse events | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Takamasa Kayama, MD, PhD, Study Chair — Yamagata University Faculty of Medicine
Locations (21):
- Japan (21):
  - Nagoya University School of Medicine, Nagoya,Showa-ku,Tsurumai-cho,65, Aichi-ken
  - Chiba University, Graduate School of Medicine, Chiba,Chuo-ku,Inohana,1-8-1, Chiba
  - Ehime University Hospital, Shitsukawa,Toon, Ehime
  - Kyushu University Hospital, Higashi-ku,Maidashi,3-1-1, Fukuoka
  - Hokkaido University Hospital, North-14 West-5 Kita-ku,Sapporo, Hokkaido
  - Nakamura Memorial Hospital, South-1,West-14,Chuou-ku,Sapporo, Hokkaido
  - Iwate Medical University, Morioka,Uchimaru,19-1, Iwate
  - St.Marianna University School of Medicine, Kawasaki,Miyamae-ku,Sugao,2-16-1, Kanagawa
  - Kumamoto University Medical School, Kumamoto,Honjo,1-1-1, Kumamoto
  - Kyoto University Hospital, Kyoto,Sakyo-ku,Syogoinkawara,54, Kyoto
  - Tohoku University Hospital, Sendai,Aoba-ku,Seiryo-machi,1-1, Miyagi
  - Niigata University Medical and Dental Hospital, Niigata,Asahimachi-dori,1-754, Niigata
  - Saitama Medical School Hospital, Iruma-gun,Moroyama-machi,Morohongo,38, Saitama
  - The University of Tokyo Hospital, Bunkyo-ku,Hongo,7-3-1, Tokyo
  - National Cancer Center Hospital, Chuo-ku,Tsukiji,5-1-1, Tokyo
  - Teikyo University School of Medicine, Itabashi-ku,Kaga,2-11-1, Tokyo
  - Kyorin University School of Medicine, Mitaka,Shinkawa,6-20-2, Tokyo
  - Tokyo Women's Medical University, Shinjuku-ku,Kawada-cho,8-1, Tokyo
  - Keio University Hospital, Shinjuku-ku,Shinanomachi,35, Tokyo
  - Yamagata University Faculty of Medicine, Yamagata City,Iida-nishi, 2-2-2, Yamagata
  - University of Yamanashi Faculty of Medicine, Nakakoma,Tamaho,Shimokato,1110, Yamanashi

REFERENCES:
- [Derived] Simeoli C, Di Paola N, Stigliano A, Lardo P, Kearney T, Mezosi E, Ghigo E, Giordano R, Mariash CN, Donegan DM, Feelders RA, Hand AL, Araque KA, Moraitis AG, Pivonello R. Relacorilant or surgery improved hemostatic markers in Cushing syndrome. J Endocrinol Invest. 2025 Mar;48(3):671-680. doi: 10.1007/s40618-024-02468-2. Epub 2024 Sep 21. PMID 39305441
- See also: Related Info — http://www.jcog.jp/